CLINICAL TRIAL: NCT06896851
Title: The Effect of Su Jok on Dysmenorrhea:Randomized Placebo-Controlled Trial
Brief Title: The Effect of Su Jok on Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Hülya Elmalı Şimşek, Assistant Proffesor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14.2024fbu
Record Dates: First submitted 2025-03-04; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea; pain; su jok
MeSH Terms: conditions — Dysmenorrhea; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Su Jok Group (Experimental): Sujok is applied with black pepper seeds to the appropriate point on the hand.
  Interventions: Other: Su Jok
- Placebo Control Group (Sham Comparator): Black pepper seeds are applied to the sham point.
  Interventions: Other: Sham point using

INTERVENTIONS:
Other: Su Jok — a type of acupressure includs hand massage
  Arms: Su Jok Group
Other: Sham point using — unrelated point using for acupressing
  Arms: Placebo Control Group

SUMMARY:
This study aims to determine the effect of Su Jok application in reducing menstrual pain.The main question it aims to answer is

-Is Su Jok practice effective in reducing the severity of dysmenorrhea? The researcher will perform a sham application to see the effect of the application.

Participants will perform the application on the first day they have pain during their 3 menstrual cycles. They will evaluate and record their pain with VAS.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles (21-35 days)
* have abdominal pain in the last three cycles
* Those who want to participate in the study as a volunteer

Exclusion Criteria:

* have any health problems that may affect the menstrual cycle (ovarian cysts, etc.
* use hormonal medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Pain assesment | " Every hour until 4 hours after the onset of pain on the first day of the cycle (each cycle is 28-35 days) and it will be for 3 cycle.
  Pain assessment is made with Visual Analog Scale(0-10 points, high score means pain severity is high) in three menstrual cycles (up to 105 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahçe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared when the research is accepted for publication.